CLINICAL TRIAL: NCT06381843
Title: A Clinical Study to Evaluate the Safety and Immunogenicity of the Recombinant COVID-19 Vaccine (Sf9 Cell) as a Booster in People Aged 18-60 Years
Brief Title: A Clinical Study to Evaluate the Safety and Immunogenicity of the Recombinant COVID-19 Vaccine (Sf9 Cell) as a Booster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WSKCT004
Record Dates: First submitted 2024-04-23; First posted 2024-04-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant COVID-19 Vaccine (Sf9 Cell) (Experimental): Participants who received 3 doses of Inactivated COVID-19 vaccines with the third dose at least 6 months (≥180 days) prior to enrolment. N=60 Intervention: Recombinant COVID-19 Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 Vaccine (Sf9 Cell)
- Inactivated COVID-19 vaccines (Active Comparator): Participants who received 3 doses of Inactivated COVID-19 vaccines with the third dose at least 6 months (≥180 days) prior to enrolment. N=60 Intervention: COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Recombinant COVID-19 Vaccine (Sf9 Cell) — 1dose, Intramuscular Injection
  Arms: Recombinant COVID-19 Vaccine (Sf9 Cell)
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — 1dose, Intramuscular Injection
  Arms: Inactivated COVID-19 vaccines

SUMMARY:
A observer-blind, randomized, controlled, investigator-initiated clinical trial to evaluate the safety and immunogenicity of a booster vaccination with Recombinant COVID-19 vaccine (Sf9 Cell) in a population aged 18-60 years old who have completed 3 doses vaccination with COVID-19 Vaccine (Vero Cell), Inactivated ≥ 6 months at least 6 months prior to enrolment. The study uses a non-inferiority design to compare between schedules with Recombinant COVID-19 Vaccine (Sf9 Cell) versus COVID-19 Vaccine (Vero Cell) Inactivated as the booster dose. Participants, laboratory and analysing statisticians will remain blind to treatment allocation.

A total of 120 participants will be enrolled, participants will be randomized 1:1 to receive a single dose of Recombinant COVID-19 vaccine (Sf9 Cell) (test group) or COVID-19 Vaccine (Vero Cell), Inactivated.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 18-60 years old, voluntarily sign the ICF approved by the ethics committee before any research procedure begins, and agree to participate in this research;
* (2) Subjects who are in line with the immunization of this product after medical history, physical examination and clinical judgment are healthy;
* (3) Participate in this clinical trial after completing 3 doses of immunization ≥ 6 months (calculated based on the date of the last vaccination as 0) in accordance with the domestically approved inactivated vaccine vaccination program, and can provide relevant vaccination certificates;
* (4) The subjects are able and willing to comply with the requirements of the clinical trial protocol, and can complete the study follow-up of about 12 months;
* (5) Males and females of childbearing age who are fertile voluntarily use effective contraceptive measures (such as condoms, intrauterine devices, spermicides) from the signing of the informed letter to 6 months after the completion of vaccination, and contraceptive use is not allowed medicine. Female subjects had a negative pregnancy test and agreed not to breastfeed during the study period and for at least 3 months after vaccination with the experimental vaccine.
* (6) Underarm body temperature <37.3℃.

Exclusion Criteria:

* (1) Positive SARS-CoV-2 RT-PCR test at screening;
* (2) A history of human coronavirus infection or disease history such as novel coronavirus (SARS-CoV-2), severe acute respiratory syndrome (SARS), and Middle East respiratory syndrome (MERS);
* (3) Those with previous medical history or family history of convulsions, epilepsy, encephalopathy or mental illness;
* (4) Persons with fainting needles;
* (5) Those who plan to become pregnant or perform sperm and egg donation during the trial period;
* (6) History of allergy or allergic reaction to any vaccine and its excipients, such as: allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, angioedema, etc.;
* (7) Have received any vaccine within 30 days before vaccination of this research vaccine or plan to receive any other vaccine other than this research vaccine during this research;
* (8) Participate in any other interventional experimental device or drug research within 30 days before screening, or are currently using other experimental drugs or within 5 half-lives after the last administration of the research drug;
* (9) Hereditary bleeding tendency or abnormal coagulation function (such as cytokine deficiency, coagulation disorder or platelet disorder), or a history of severe bleeding, or a history of massive bleeding or ecchymosis after intramuscular injection or venipuncture;
* (10) According to known medical history or diagnosis, it is confirmed to have diseases that affect the function of the immune system, including cancer, congenital or acquired immunodeficiency (eg: human immunodeficiency virus (HIV) infection), uncontrolled autoimmune diseases;
* (11) There are serious or uncontrollable diseases of the respiratory system, cardiovascular diseases, nervous system diseases, blood and lymphatic system diseases, liver and kidney diseases, metabolic and skeletal diseases that are judged by the investigator to affect the evaluation of the results of this study;
* (12) Asplenia or functional asplenia;
* (13) Long-term use (≥14 days of continuous use) of immunosuppressive drugs or other immunomodulatory drugs (such as corticosteroids: prednisone or similar drugs) within 6 months before the vaccine for this trial, but topical drugs are allowed ( Such as ointment, eye drops, inhalation or nasal spray), topical application should not exceed the dose recommended in the instructions or have any signs of systemic exposure;
* (14) Received immunoglobulin and/or blood products within 3 months before the vaccine for this trial;
* (15) Patients undergoing anti-tuberculosis treatment;
* (16) According to the judgment of the investigator, due to various medical, psychological, social or other conditions, it is contrary to the experimental protocol, or affects the subject's signing of informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | Day 0-30 post-boost dose.
Geometric mean titer (GMT) of specific neutralizing antibody against SARS-CoV-2 prototype strain | Day 30 post-boost dose.
Geometric mean titer (GMT) of specific neutralizing antibody against SARS-CoV-2 Omicron variant | Day 30 post-boost dose.

SECONDARY OUTCOMES:
Geometric mean increase (GMI) of specific neutralizing antibody against SARS-CoV-2 prototype strain | Day 30 post-boost dose.
Geometric mean increase (GMI) of specific neutralizing antibody against SARS-CoV-2 Omicron variant | Day 30 post-boost dose.
GMT and GMI of specific neutralizing antibody against SARS-CoV-2 prototype strain | Day 7, day 14, month 3 and month 6 after the booster dose.
GMT and GMI of specific neutralizing antibody against SARS-CoV-2 omicron variant | Day 7, day 14, month 3 and month 6 after the booster dose.
GMT and GMI of IgG antibodies against SARS-CoV-2 S protein RBD | Day 7, day 14, day 30, month 3 and month 6 after the booster dose.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided